CLINICAL TRIAL: NCT05180110
Title: A Performance Evaluation of the LumiraDx Point of Care CRP Assay.
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00008
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Inflammation; Infections; Tissue Injury
MeSH Terms: conditions — Inflammation; Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: IVD Performance Evaluation Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symptoms of inflammation, Infection, tissue injury (Experimental): Venous blood draw of up to 24mL and up to 6 capillary fingersticks
  Interventions: Diagnostic Test: Venepuncture; Diagnostic Test: Fingerstick

INTERVENTIONS:
Diagnostic Test: Venepuncture — Venous blood draw
Diagnostic Test: Fingerstick — Capillary blood draw

SUMMARY:
In patients with symptoms of infection, tissue injury and inflammatory disorders the study will evaluate agreement between the CRP measurements from the LumiraDx POC CRP assay and the Siemens Dimension Xpand Plus CRP assay, as an aid in evaluation and detection of infection, tissue injury and inflammatory disorders.

DETAILED DESCRIPTION:
This is a performance evaluation study designed to assess the precision and accuracy of the LumiraDx point of Care (POC) C-reactive Protein (CRP) test when used in patients presenting with symptoms of infection, tissue injury or inflammatory disorder.

The LumiraDx POC CRP test is a quantitative immunoassay providing results in under 10 minutes. The accuracy of the LumiraDx POC CRP test will be assessed using capillary whole blood, venous blood, and plasma samples, by comparison to the CRP results obtained from the same individuals as analysed by trained laboratory professionals using the reference device, Siemens Dimension Xpand Plus CRP assay. The results of this study are intended to be used for regulatory filings for use as an in vitro diagnostic test in the UK, European Union (EU) and other relevant geographies.

Adults (aged 18 and over at time of consent) presenting to the study sites with symptoms of infection, tissue injury or inflammatory disorder will be included in the study. Approximately 250 patients will be recruited to ensure that sufficient suitable patients are enrolled and to allow for a small level of exclusions.

After obtaining informed consent, blood tube samples will be drawn and fingerstick samples of capillary blood will be taken from the subject, these will be applied directly onto unique test strips for immediate measurement of CRP on the LumiraDx POC instrument.

The CRP results obtained via the LumiraDx CRP test will be used in a set of comparative analyses designed to determine the performance characteristics of the test. This study is an observational, cross-sectional design. As an observational study of an investigative device, results obtained during the course of the study will not inform or alter patient management or treatment decisions in any way.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and over at the time of consent
* Willing and able to provide written informed consent and comply with study procedures
* Presenting with symptoms of infection, tissue injury, inflammatory disorders. This includes but not limited to : respiratory tract infection (upper and lower), rheumatoid arthritis, Lupus, burns, trauma, inflammatory bowel disease.

Exclusion Criteria:

* The patient is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic or drug including either treatment or therapy.
* Skin lesions or conditions that would preclude a fingerstick and/or a venous blood draw.
* Patient has previously participated in this study
* Any patient with critical illness or requiring a time critical intervention
* Patient with end of life or palliative care
* Patient suffering from the following conditions: Myeloma, monoclonal gammopathy, extreme lipaemia
* Patient is deemed medically unfit to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
To determine the performance of the LumiraDx POC CRP assay when compared to the Siemens Dimension Xpand Plus CRP in patients with symptoms of infection, inflammation, or injury. | 2 months
  Measurement of blood samples from patients with symptoms of inflammation, infection or injury in a reference method and in the LumiraDx method to assess accuracy of the LumiraDx method

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Gray, MD, Principal Investigator — NHS Lothian; James Harnett, Principal Investigator — University College London Hospital NHS Foundation Trust; Phil Moss, Principal Investigator — St Georges University Hospitals NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Royal Infirmary Edinburgh, Edinburgh
  - St Georges Hospital, London
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No